CLINICAL TRIAL: NCT02997085
Title: Virtual Reality for Pain Management Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Seton Healthcare Family (Other)
Responsible Party: Principal Investigator, Mark B. Powers, Research Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-09-0140
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Pain, Acute
Keywords: Pain; Virtual Reality; Opioid; Prescription pain reliever; Treatment
MeSH Terms: conditions — Acute Pain; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Live-Action 360° Video Virtual Reality (Experimental)
  Interventions: Device: Live-Action 360° Video Virtual Reality
- CGI 360° Video Virtual Reality (Active Comparator)
  Interventions: Device: CGI 360° Video Virtual Reality
- Waitlist (No Intervention): Participants randomized to the waitlist group will complete all study procedures except the VR exposure. After completion of the study visit, participants in the waitlist condition will be given the option of viewing either the Live-Action 360° 3D HD VVR or the CGI 360° 3D VVR.

INTERVENTIONS:
Device: Live-Action 360° Video Virtual Reality — 360° Video Virtual Reality (VVR) is made by filming with multiple HD cameras carefully arranged to capture all angles in a 360° area of a live action event. Then those angles are stitched together in post-production into a 360-degree texture sphere and the sphere is then mapped to the head tracker on the users head mounted display (HMD). Leading to the effect that when a user turns his head, the user's view of the live action video footage turns with them in real time allowing the user to look around anywhere in the 360 degrees of filmed footage of the live action event. Participants randomized to the Live-Action 360° VVR group will be outfitted with a Samsung Gear VR HMD and will view a 9-minute live-action 360° VVR video. The 9 minutes of footage will be alternating 30 second clips of central Texas locations.
  Arms: Live-Action 360° Video Virtual Reality
Device: CGI 360° Video Virtual Reality — Participants randomized to the CGI 360° VVR condition will also be outfitted with a Samsung Gear VR head mounted display. Participants will view the same content for the same duration as in the Live-Action 360° VVR condition, but the footage will be animated instead of live-action footage.
  Arms: CGI 360° Video Virtual Reality

SUMMARY:
Virtual Reality (VR) is one non-pharmacological method that has shown promise as an effective means of decreasing pain levels following treatment, and for significant periods of time. Additionally, neurobiology studies of VR have demonstrated a decrease in brain activity associated with pain. While VR is clearly a promising, drug-free option for pain treatment, existing VR systems are expensive and use unconvincing graphics. Recent advances in VR technology (i.e., improved realism and immersion using 360-degree 3D technology and more affordable delivery systems) allow the development of more realistic and more cost-effective applications. Capitalizing on these advances and the investigators' experiences with VR intervention development and evaluation, the current study will test a state-of-the-art VR experience in pain management intervention (Live-Action 360° Video Virtual Reality(VVR)) and compare it to established standard computer generated imagery (CGI) 360° VVR content for pain management intervention in a medical setting. The participant's participation will help the investigators determine which VR intervention is most effective in reducing acute pain in hospital patients.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65
* Reports experiencing current pain not typical of day-to-day experience during Pre-Treatment Pain Questionnaire at the onset of study visit by answering "Yes" to the first question of the questionnaire. There is no specific threshold of how much pain the participant must be in to be eligible for this study. The participant must be experiencing current pain that is not related to day-to-day, normal experiences (such as minor headaches, sprains, and toothaches).
* Scores a 15 on the Glasgow Coma Scale and a 7 or above on the abbreviated Mini Mental Status Exam.
* Patient in the acute and critical palliative care units, post surgical units, or acute care orthopedic units at University Medical Center Brackenridge in Austin, TX.
* Willing and able to provide informed consent and participate in the study visit and study follow-up questionnaire.

Exclusion Criteria:

* Hearing or visually impaired where participant cannot use the Samsung Gear VR.
* Does not report experiencing current pain during Pre-Treatment Pain Questionnaire at the onset of study visit.
* Scores below a 15 on the Glasgow Coma Scale and/or below a 7 on the abbreviated Mini Mental Status Exam
* Limited mental competency and the inability to give informed, voluntary, written consent to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Powers, Ph.D., Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Live-Action 360° Video Virtual Reality | CGI 360° Video Virtual Reality | Waitlist
Started | 34 | 35 | 34
Completed | 34 | 35 | 34
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Live-Action 360° Video Virtual Reality | CGI 360° Video Virtual Reality | Waitlist | Total
Number analyzed (Participants) | 34 | 35 | 34 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 34 | 31 | 96
  >=65 years | 3 | 1 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.03 (14.14) | 43.83 (13.51) | 44.62 (16.17) | 43.17 (14.58)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 18 | 12 | 11 | 41
  Male | 16 | 23 | 22 | 61
  Prefer Not to Report | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 6 | 20
  Not Hispanic or Latino | 27 | 28 | 28 | 83
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 6 | 14
  White | 27 | 29 | 28 | 84
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 34 | 35 | 34 | 103
Pain Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Pain Questionnaire was used to assess the participant's pain prior to receiving VR treatment, following VR treatment, and at the ten-minute follow-up assessment. It was derived from the Brief Pain Inventory (BPI) and contains the Numerical Rating Scales (NRS) to assess the participant's pain as outlined by recommendations for outcome measures in clinical pain trials.The NRS was also chosen because it could be administered orally if patients could not use their hands to write or use the iPad. Scores start at 0 being no pain at all and 10 being pain as bad as you can imagine. Pain is current
  units on a scale | 5.97 (1.88) | 5.22 (2.02) | 6.29 (2.37) | 5.83 (2.27)
Present Mood Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Present Mood Questionnaire was used to assess the participant's current mood. The survey uses a labeled (0-10) NRS to measure the extent to which the participant feels sad, anxious, happy, and tranquil. It was administered at each of the three assessments (baseline, post-treatment, follow-up) except for in waitlist participants, for whom it was not administered at the final assessment to reduce participant burden. Higher values indicate worse outcomes for depression and anxiety and better outcomes for happiness and tranquility.
  units on a scale
    Depression | 2.62 (3) | 2.17 (2.71) | 2.15 (2.35) | 2.33 (2.68)
    Anxiety | 4 (3.47) | 2.86 (3.05) | 3.18 (3.33) | 3.37 (3.29)
    Happy | 4.12 (3.22) | 4.71 (3.27) | 5.62 (3.58) | 4.80 (3.40)
    Tranquil | 5.44 (3.25) | 6.06 (2.78) | 6.21 (2.71) | 5.86 (2.89)

OUTCOME MEASURES:

1. Primary Outcome: Post-Treatment Pain Questionnaire
Description: The Pain Questionnaire was used to assess the participant's pain prior to receiving VR treatment, following VR treatment, and at the ten-minute follow-up assessment. It was derived from the Brief Pain Inventory (BPI) and contains the Numerical Rating Scales (NRS) to assess the participant's pain as outlined by recommendations for outcome measures in clinical pain trials.The NRS was also chosen because it could be administered orally if patients could not use their hands to write or use the iPad. Scores start at 0 being no pain at all and 10 being pain as bad as you can imagine. Pain is current
Time Frame: Immediately following intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Live-Action 360° Video Virtual Reality | CGI 360° Video Virtual Reality | Waitlist
Number analyzed (Participants) | 34 | 35 | 34
score on a scale | 3.03 (2.3) | 2.77 (2.13) | 6.37 (2.23)

2. Secondary Outcome: Follow-Up Pain Questionnaire
Description: as for outcome 1
Time Frame: Every 10 minutes for 40 minutes following intervention and 1 week following intervention. Meaned.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Live-Action 360° Video Virtual Reality | CGI 360° Video Virtual Reality | Waitlist
Number analyzed (Participants) | 34 | 35 | 34
units on a scale | 4.2 (2.32) | 4.14 (2.72) | 3.7 (3.04)

3. Secondary Outcome: Presence Inventory
Description: Self-report measure that assesses the degree of spatial presence, involvement, ecological validity, overall presence, and negative effects experienced during the VR intervention. Questions are asked on a scale of 0-10 with 0 being strongly Disagree and 10 being strongly agree. Spatial presence has a total of 3 questions for a total score of 30, and higher values mean increased spatial prescence. Ecological Validity has a total of 4 questions for a total score of 40 and higher values mean increased ecological validity. Higher for these two subscales indicate a better outcome. Negative Effects has a total of 4 questions for a total score of 40, and higher values mean more negative effects. Higher scores for this subscale indicate a worse outcome. Questions on the scale are summed.
Time Frame: Immediately following intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Live-Action 360° Video Virtual Reality | CGI 360° Video Virtual Reality
Number analyzed (Participants) | 34 | 35
units on a scale
  Ecological Validity | 35.06 (7.69) | 25.62 (12.09)
  Spatial Presence | 25.79 (6.99) | 22.18 (8.97)
  Negative Effects | 1.09 (2.23) | 2 (5.68)

4. Secondary Outcome: Absorption Survey
Description: Self-report measure that assesses participant engagement with the virtual world. Questions are asked on a scale of 0-10 with 0 being strongly Disagree and 10 being strongly agree. There are 12 questions with a total score of 120. Higher scores indicate a better outcome and increased participant engagement.
Time Frame: Immediately after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Live-Action 360° Video Virtual Reality | CGI 360° Video Virtual Reality
Number analyzed (Participants) | 34 | 35
units on a scale | 104.32 (16.52) | 96.2 (18.34)

5. Secondary Outcome: Present Mood Questionnaire
Description: The Present Mood Questionnaire was used to assess the participant's current mood. The survey uses a labeled (0-10) NRS to measure the extent to which the participant feels sad, anxious, happy, and tranquil. It was administered at each of the three assessments (baseline, post-treatment, follow-up) except for in waitlist participants, for whom it was not administered at the final assessment to reduce participant burden. Higher values indicate worse outcomes for depression and anxiety and better outcomes for happiness and tranquility.
Time Frame: Every 10 minutes for 40 minutes following intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Live-Action 360° Video Virtual Reality | CGI 360° Video Virtual Reality | Waitlist
Number analyzed (Participants) | 34 | 35 | 34
units on a scale
  Depression | .7 (1.45) | .85 (1.88) | 2.25 (3.13)
  Anxiety | 1.24 (3.18) | 1.21 (2.27) | 2.25 (2.76)
  Happy | 6.52 (2.54) | 6.24 (3.38) | 5.34 (3.39)
  Tranquil | 7.7 (2.3) | 7.62 (2.71) | 6.56 (2.65)

6. Secondary Outcome: Attitudes Toward the Experience Survey
Description: Self-report measure that assesses the participant's attitude toward the VR experience. Questions are asked on a scale of 0-10 with 0 being strongly Disagree and 10 being strongly agree. There are 12 questions for a total score of 120. Higher scores mean a more positive attitude towards the experience and is a better outcome.
Time Frame: Immediately after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Live-Action 360° Video Virtual Reality | CGI 360° Video Virtual Reality
Number analyzed (Participants) | 34 | 35
units on a scale | 74.35 (10.93) | 67.51 (16.49)

ADVERSE EVENTS:
Time Frame: One year
Description: Waitlist group was enrolled in other groups after the wait. Their numbers are included in the other group's counts. Participants in waitilist chose their own groups so numbers are not even.
Arm/Group | Live-Action 360° Video Virtual Reality | CGI 360° Video Virtual Reality
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/37
Other Adverse Events (participants affected / at risk) | 9/66 | 7/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Live-Action 360° Video Virtual Reality (N=66) | CGI 360° Video Virtual Reality (N=37)
Eyestrain (Eye disorders) | 6 (6) | 5 (5)
Dizzy (Nervous system disorders) | 4 (4) | 4 (4) — Just dizzy from device.
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) — Nausea from device usage.
Headache (Nervous system disorders) | 2 (2) | 2 (2) — Headache from device usage

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2014-10-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT02997085/Prot_000.pdf